CLINICAL TRIAL: NCT05344963
Title: Deformation Imaging by Strain in Chronic Heart Failure Over Gliflozins: an Echocardiographic Register on Sodium-GLucose coTransporter-2 Inhibitors
Acronym: DISCOVERSGLT2i
Status: Completed | Type: Observational
Sponsor: Matteo Cameli (Other)
Collaborators: Fondazione Toscana G. Monasterio, Pisa (Unknown); University Of Perugia (Other); Section of Cardiology, Department of Medicine, University of Verona, Verona (Unknown); Department of Cardiovascular and Thoracic Sciences, Fondazione Policlinico Universitario A. Gemelli, IRCCS, Università Cattolica del Sacro Cuore, Rome (Unknown); Cardiology and Arrhythmology Clinic, Marche Polytechnic University, 60121 Ancona (Unknown); Cardiology Department, Ospedale Guglielmo da Saliceto - Piacenza (Unknown); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); ProMISE, University Hospital Paolo Giaccone, University of Palermo (Unknown); Department of Cardiovascular Disease - AUSL Romagna, Division of Cardiology, Ospedale S. Maria Delle Croci, Viale Randi 5, 48121, Ravenna (Unknown); Department of Medical and Surgical Specialties, Radiological Sciences and Public Health, University of Brescia, Brescia (Unknown); Department of Biomedical Sciences for Health, University of Milano, Milan (Unknown); Division, of Cardiology, 'A. De Gasperis' Cardio Center, ASST Grande Ospedale Metropolitano Niguarda, Piazza Ospedale Maggiore 3, 20162, Milan (Unknown); Department of Advanced Biomedical Science, Federico II University Hospital, Naples (Unknown); Department of Thoracic, Heart and Vascular Diseases, Maggiore della Carità Hospital, Novara (Unknown); Divisione di Cardiologia, Ospedale S. Maria del Carmine, Rovereto, TN (Unknown); ASST-Rhodense; Ospedale di Circolo di Rho (Unknown); Cardio-Thoracic-Vascular Department. University Hospital San Giovanni di Dio e Ruggi d'Aragona. Salerno (Unknown); Centro Medico Sant'Agostino, Milano (Unknown); Università Politecnica delle Marche, Ospedali riuniti di Ancona (Unknown); Department of Cardiology, Policlinico Universitario Campus Bio-Medico, Via Álvaro del Portillo, 21, Roma (Unknown)
Responsible Party: Sponsor-Investigator, Matteo Cameli, Professor, Azienda Ospedaliera Universitaria Senese
Organization: Azienda Ospedaliera Universitaria Senese (Other)
Other Study IDs: DISCOVER SGLT2i
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Sodium-GLucose coTransporter-2 Inhibitors; Heart Failure With Reduced Ejection Fraction
Keywords: Echocardigraphy; Speckle tracking; Strain; SGLT2i
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Sodium-GLucose coTransporter-2 inhibitors — Evaluation of the modification of conventional and advanced echocardiographic parameters, focusing on speckle tracking and three-dimensional echocardiography (optional), in patients with HFrEF after treatment with the SGLT2i drugs Dapagliflozin and Empagliflozin

SUMMARY:
It is an observational, cohort, prospective, multicentre, Italian, non-profit study, with the aim of evaluating the modification of conventional and advanced echocardiographic parameters, focusing on speckle tracking and three-dimensional echocardiography (optional), in patients with HFrEF after treatment with SGLT2i Dapagliflozin and Empagliflozin.

Participation in the study will last for approximately 18 months, and a total of 300 patients will be enrolled at the various Research Centers.

The enrolled patients will undergo a first evaluation in which the anamnestic, clinical and conventional and advanced echocardiographic data will be recorded. At this point, the patient will start SGLT2i.

After starting SGLT2i, a second evaluation will be carried out with a cardiological visit at 6 months, in which the same data listed above will then be recorded.

At the end of the evaluation, the clinical follow-up will be continued for the duration of 1 year, in number and frequency according to clinical indication.

ELIGIBILITY:
Inclusion Criteria:

1. Providing informed consent prior to any specific study procedure
2. Female or male outpatient patients > 18 years
3. Have heart failure and left ventricular ejection fraction <= 40%, according to the ESC definition
4. Already on therapy with an angiotensin converting enzyme (ACE) inhibitor or sacubitril / valsartan, a beta-blocker and mineralocorticoid receptor antagonist (MRA) and be initiated for treatment with SGLT2i for therapy optimization

Exclusion Criteria:

1. Involvement in study planning and / or conducting (applies to both investigator staff and study site staff)
2. Age <18 years
3. For women only - ongoing pregnancy (confirmed with positive pregnancy test)
4. For women only - breastfeeding
5. Poor quality of echocardiographic images which compromises a correct speckle tracking analysis
6. Failure to sign informed consent.
7. Previous treatment with SGLT2i.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with heart failure and EF <= 40% and already on an ACE inhibitor / angiotensin-neprilysin receptor (ARNI) inhibitor, a beta blocker and an aldosterone receptor inhibitor, where treatment will be initiated with SGLT2i for optimization of therapy for heart failure, according to the latest ESC guidelines.
Sampling Method: Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Predictors of remodeling and improvement in LV systolic and diastolic function | 18 months
  A univariate and multivariate logistic regression analysis will be performed to search for predictors of remodeling and improvement in LV systolic and diastolic function at 6 months, with particular attention to advanced echocardiography parameters.

SECONDARY OUTCOMES:
Combined outcome 12 months from the third evaluation (18 months from the start of therapy) including death from cardiovascular causes, appropriate defibrillator discharge, hospitalizations or episodes of atrial fibrillation. | 18 months
  Uni and multivariate Cox analyzes will be performed for predictors of cardiovascular events and the quality of the model will then be estimated by time-dependent ROC analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Diagnostica Cardiovascolare, AOU Senese Policlinico Le Scotte, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Result] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829